CLINICAL TRIAL: NCT01391832
Title: Novel Treatment of Emotional Dysfunction in PTSD
Brief Title: Novel Treatment of Emotional Dysfunction in Post Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, John Hart, Jr., Professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 092010-035
Record Dates: First submitted 2011-07-05; First posted 2011-07-12 (Estimated); Results first posted 2020-10-01 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Post Traumatic Stress Disorder
Keywords: rTMS; PTSD; Post Traumatic Stress Disorder; repetitive transcranial magnetic stimulation; combat related PTSD; OEF; OIF; Veterans; operation enduring freedom; operation iraqi freedom; CPT; cognitive processing therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Transcranial Magnetic Stimulation; 2-cyclohexylidenhydrazo-4-phenyl-thiazole; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sham rTMS (Sham Comparator): Sham Treatment Intervention: Device: Repetitive Transcranial Magnet Stimulation (sham treatment)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Behavioral: Cognitive Processing Therapy
- active rTMS (Active Comparator): Active Repetitive Transcranial Magnet Stimulation treatment
  Intervention: Device: Active rTMS of dorsolateral pre-frontal cortex
  Interventions: Behavioral: Cognitive Processing Therapy; Device: Repetitive Transcranial Magnet Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — For the sham rTMS with CPT group, the rTMS coil will be placed over the right prefrontal scalp region with the MagStim Rapid Stimulator set to the sham mode so that all conditions are similar to the active delivery mode except that transcranial magnetic stimulation is not administered to the scalp and does not down modulate the right frontal lobe.
  Other Names: rTMS; magnet stimulation
  Arms: Sham rTMS
Behavioral: Cognitive Processing Therapy — Cognitive Processing Therapy (CPT) is a 12 session evidenced based, trauma-focused treatment for PTSD. CPT is a cognitive therapy based on information processing theory and includes components which help the client to (a) access her or his memory of the event, (b) identify and experience her or his emotions until they have been extinguished, and (c) identify and challenge beliefs about the event itself and beliefs about self and the world which have been altered because of the combat related trauma.
  Other Names: CPT; behavioral training; behavioral therapy
Device: Repetitive Transcranial Magnet Stimulation (rTMS) — For the active rTMS with CPT group, the rTMS coil will be placed over the right prefrontal scalp region with the MagStim Rapid Stimulator set to the active mode. After motor threshold determination, the stimulator coil is positioned over the dorsolateral prefrontal cortex - DLPFC (Brodmann Area 9/46). The right frontal rTMS will safely, reversibly, and temporarily down modulate the right frontal lobe. The conducting coil is placed over the scalp while electrical current pulses pass through the coil. This alternating current turned on and off rapidly produces magnetic pulses (1.5-2.0 Tesla strength) that last for 100 - 300 microseconds. The time-varying magnetic pulses induce an electrical field that will result in current flow in neural tissue, thereby activating or deactivating cortex subjacent to the coil.
  Arms: active rTMS

SUMMARY:
The objective will be to determine if adding repetitive transcranial magnetic stimulation prior to Cognitive Processing Therapy significantly enhances recovery from hyperarousal symptoms in individuals with combat related post traumatic stress disorder and improves clinical outcome.

The investigators have assembled a multimodal human performance laboratory including 64 channel EEG and repetitive transcranial magnetic stimulation system. These resources combined with the neuroimaging capabilities of the Advanced Imaging Research Center (AIRC) at UT Southwestern and skilled Cognitive Processing Therapy (CPT) practitioners will be used in this study.

The study involves approximately 19 visits. Treatment is once a week for 12 weeks followed by a 1 month, 3 month and 6 month follow-up appointments.

DETAILED DESCRIPTION:
We will first screen participants between the ages of 18 and 60 years for symptoms of PTSD as determined by subjective reporting. We will also screen for healthy control participants to participate in comparison assessment phases of the study. After meeting pre-screen criteria, a more extensive screening to determine the eligibility of each subject will be performed. This will be followed by an EEG. The EEG system measures event-related potentials (ERPs), which explain certain cognitive processes based on changes in the amplitude and timing of electrical changes recorded from the surface of the scalp. We will use an ERP task that includes combat-threatening stimuli as the novel oddball probe to assess P300 response. The amplitude of the P300 (positive amplitude recorded 300 milliseconds after stimulus onset) is used to differentiate between hypo-, normo-, and hyper-arousability. Identifying those with hyperarousal on P300 response on ERP allows for identification of PTSD patients with subjective and objective measures of hyperarousal. The participants will then be scheduled for a neuroimaging session. During neuroimaging, participants will have structural and functional brain scans acquired, including a functional MRI scan using the same threatening/nonthreatening stimuli, thus providing another objective measure of hyperarousal.

Participants will then have active or sham 1 Hz repetitive transcranial magnetic stimulation (rTMS) administered to the right frontal lobe as well as Cognitive Processing Therapy (CPT) once per week for twelve weeks (total 12 rTMS-CPT sessions). Studies have shown that rTMS applied externally to the forehead in the region of the dorsal lateral forehead will safely, reversibly, and painlessly down-modulate the frontal lobe on the side of the head to which it is applied. Our preliminary studies have shown that application of frontal rTMS can reduce the response to threatening stimuli temporarily and this can optimize the effectiveness of the CPT. Following the 12 sessions of rTMS-CPT, the EEG and neuroimaging will be repeated to test for changes in brain function.

In summary, the study involves approximately 19 visits. Treatment is once a week for 12 weeks followed by a 1 month, 3 month and 6 month follow-up appointments.

* The first 2-3 visits involve an informed consent, a baseline assessment, EEG and neuroimaging.
* Visits 4-15 are the rTMS/CPT sessions.
* Visit 16 is a 1 month follow-up, post-treatment assessment and EEG.
* Visit 17 is a post-treatment neuroimaging visit.
* Visit 18 is the 3 month follow up assessment.
* Visit 19 is the 6 month follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Veterans of Operation Iraqi Freedom (OIF) or Operation Enduring Freedom (OEF)
* 18-60 years
* Diagnosis or symptoms of Combat related PTSD/ PCL Score Indicative of diagnosis (prior diagnosis not required).
* English speaking
* Participants will be screened for exclusionary medical and mental health history.

This study is also looking for civilian and miltary control subjects for assessment phase participation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2011-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Hart Jr., M.D., Principal Investigator — The University of Texas at Dallas; F. Andrew Kozel, M.D., Study Director — University of Texas
Locations (1):
- University of Texas at Dallas, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans previously deployed to combat regions from 2001 to present (e.g., Operation Enduring Freedom (OEF), Operation Iraq Freedom (OIF), and Operation New Dawn (OND) with current combat-related PTSD symptoms were recruited from the community.
Groups:
- Sham rTMS: Sham Treatment Intervention: Device: Repetitive Transcranial Magnet Stimulation (sham treatment)
  Repetitive Transcranial Magnetic Stimulation (rTMS): For the sham rTMS with CPT group, the rTMS coil will be placed over the right prefrontal scalp region with the MagStim Rapid Stimulator set to the sham mode so that all conditions are similar to the active delivery mode except that transcranial magnetic stimulation is not administered to the scalp and does not down modulate the right frontal lobe.
  Cognitive Processing Therapy (CPT): CPT is a 12 session evidenced based, trauma-focused treatment for PTSD. CPT is a cognitive therapy based on information processing theory and includes components which help the client to (a) access her or his memory of the event, (b) identify and experience her or his emotions until they have been extinguished, and (c) identify and challenge beliefs about the event itself and beliefs about self and the world which have been alte
- Active rTMS: Active Repetitive Transcranial Magnet Stimulation treatment
  Intervention: Device: Active rTMS of dorsolateral pre-frontal cortex
  Cognitive Processing Therapy (CPT): CPT is a 12 session evidenced based, trauma-focused treatment for PTSD. CPT is a cognitive therapy based on information processing theory and includes components which help the client to (a) access her or his memory of the event, (b) identify and experience her or his emotions until they have been extinguished, and (c) identify and challenge beliefs about the event itself and beliefs about self and the world which have been altered because of the combat related trauma.
  Repetitive Transcranial Magnet Stimulation (rTMS): For the active rTMS with CPT group, the rTMS coil will be placed over the right prefrontal scalp region with the MagStim Rapid Stimulator set to the active mode. After motor threshold determination, the stimulator coil is positioned over the dorsolateral prefrontal cortex - D
Period: Overall Study
Arm/Group | Sham rTMS | Active rTMS
Started | 49 | 54
1 Month Follow-Up | 30 | 31
3 Month Follow-Up | 28 | 29
Completed | 28 | 31
Not Completed | 21 | 23
Not completed — Withdrawal by Subject | 21 | 22
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Veterans previously deployed to combat regions from 2001 to present (e.g., Operation Enduring Freedom (OEF), Operation Iraq Freedom (OIF), and Operation New Dawn (OND) with current combat-related PTSD symptoms were recruited from the community.
Groups:
- Sham rTMS: Sham Treatment Intervention: Device: Repetitive Transcranial Magnet Stimulation (sham treatment)
  Repetitive Transcranial Magnetic Stimulation (rTMS): For the sham rTMS with CPT group, the rTMS coil will be placed over the right prefrontal scalp region with the MagStim Rapid Stimulator set to the sham mode so that all conditions are similar to the active delivery mode except that transcranial magnetic stimulation is not administered to the scalp and does not down modulate the right frontal lobe.
  Cognitive Processing Therapy (CPT): CPT is a 12 session evidenced based, trauma-focused treatment for PTSD. CPT is a cognitive therapy and includes components which help the client to (a) access her or his memory of the event, (b) identify and experience her or his emotions until they have been extinguished, and (c) identify and challenge beliefs about the event itself and beliefs about self and the world which have been altered because of the combat related trauma.
- Active rTMS: Active Repetitive Transcranial Magnet Stimulation treatment
  Intervention: Device: Active rTMS of dorsolateral pre-frontal cortex
  Cognitive Processing Therapy (CPT): CPT is a 12 session evidenced based, trauma-focused treatment for PTSD. CPT is a cognitive therapy and includes components which help the client to (a) access her or his memory of the event, (b) identify and experience her or his emotions until they have been extinguished, and (c) identify and challenge beliefs about the event itself and beliefs about self and the world which have been altered because of the combat related trauma.
  Repetitive Transcranial Magnet Stimulation (rTMS): For the active rTMS with CPT group, the rTMS coil was be placed over over the dorsolateral prefrontal cortex - DLPFC (Brodmann Area 9/46) and stimulation provided at 1 Hz (1.5-2.0 Tesla strength, 100 - 300 microseconds.
- Total: Total of all reporting groups
Arm/Group | Sham rTMS | Active rTMS | Total
Number analyzed (Participants) | 49 | 54 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.39 (6.13) | 32.89 (7.60) | 32.65 (6.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 44 | 53 | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 13 | 22
  Not Hispanic or Latino | 40 | 41 | 81
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 42 | 42 | 84
  African American | 6 | 7 | 13
  Other | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  United States | 49 | 54 | 103

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Follow-up in Clinician Administered Post-Traumatic Stress Disorder Scale Total Severity Score
Description: The primary outcome measure of treatment efficacy for post-traumatic stress disorder (PTSD) will be change in the Clinician Administered Post-Traumatic Stress Disorder Scale (CAPS) Total Severity Score (i.e., summed across frequency and intensity ratings for the 17 PTSD assessment items) from baseline at 1-month post-treatment. CAPS Total Severity Score ranges from 0 to 136. Difference scores were calculated as the outcome score minus the baseline score, with negative scores indicating a reduction in symptom severity from baseline (i.e., a positive treatment outcome), and differences between treatment groups in change scores were evaluated using t-tests.
Time Frame: Outcome measures will be measured as change from baseline at 1-, 3-, and 6-month follow-ups
Population: Veterans previously deployed to combat regions from 2001 to present (e.g., Operation Enduring Freedom (OEF), Operation Iraq Freedom (OIF), and Operation New Dawn (OND)) with current combat-related PTSD symptoms were recruited from the community. 103 were enrolled and randomly assigned to the treatment arms on a parallel 1:1 basis.
Measure: Mean (Standard Error); unit: change in scale score from baseline
Groups:
- Sham rTMS: Sham Treatment Intervention: Device: Repetitive Transcranial Magnet Stimulation (sham treatment)
  The rTMS coil will be placed over the right prefrontal scalp region, simulating targeting DLPFC (Brodmann Area 9/46), with the MagStim Rapid Stimulator set to the sham mode so that all conditions are similar to the active delivery mode except that transcranial magnetic stimulation is not administered to the scalp.
  Cognitive Processing Therapy (CPT): CPT is a 12 session evidenced based, trauma-focused treatment for PTSD. CPT is a cognitive therapy based on information processing theory and includes components which help the client to (a) access memory of the traumatic event, (b) identify and experience her or his emotions until they have been extinguished, and (c) identify and challenge beliefs about the event itself, about self and the world which have been altered.
- Active rTMS: Active Repetitive Transcranial Magnet Stimulation treatment
  Intervention: Device: Active rTMS of dorsolateral pre-frontal cortex The rTMS coil will be placed over the right prefrontal scalp region, targeting DLPFC (Brodmann Area 9/46), with the MagStim Rapid Stimulator set to the active mode. Alternating current turned on and off rapidly produces magnetic pulses (1.5-2.0 Tesla strength) that last for 100 - 300 microseconds (1 HZ at 110% of motor-threshold).
  Cognitive Processing Therapy (CPT): CPT is a 12 session evidenced based, trauma-focused treatment for PTSD. CPT is a cognitive therapy based on information processing theory and includes components which help the client to (a) access memory of the traumatic event, (b) identify and experience her or his emotions until they have been extinguished, and (c) identify and challenge beliefs about the event itself, about self and the world which have been altered.
Arm/Group | Sham rTMS | Active rTMS
Number analyzed (Participants) | 49 | 54
change in scale score from baseline
  1 month change from baseline: number analyzed (Participants) | 30 | 31
  1 month change from baseline | -35.59 (4.22) | -44.164 (3.8226)
  3 month change from baseline: number analyzed (Participants) | 28 | 29
  3 month change from baseline | -33.19 (4.24) | -44.95 (3.85)
  6 month change from baseline: number analyzed (Participants) | 28 | 29
  6 month change from baseline | -36.31 (4.24) | -47.76 (3.82)
Statistical Analysis 1: Comparison: Sham rTMS vs Active rTMS; Restricted maximum likelihood estimators (ReML) of the variance components were used to compute the maximum likelihood estimators of the fixed effects parameters (i.e., group, time, therapist, all two-way interaction terms, and the three-way interaction term). Thus, we did not exclude participants with missing time points; Test type: Superiority — Comparison of differences between rTMS+CPT and sham+CPT groups in change Clinical Administered Post-Traumatic Scale Total Severity Scores from baseline to 1-month follow-up; p > 0.05, Mixed Models Analysis — Predicted effects on symptom reduction were evaluated with α = 0.05 for one-tailed t-distributions, recommended for designs examining efficacy of therapeutic interventions (Overall, 1991); Restricted maximum likelihood estimators of variance components for fixed effects; Satterthwaite estimates of effective degrees of freedom; t-value on group differences in change = -1.51 — degrees of freedom = 327
Statistical Analysis 2: Comparison: Sham rTMS vs Active rTMS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Comparison of differences between rTMS+CPT and sham+CPT groups in change Clinical Administered Post-Traumatic Scale Total Severity Scores from baseline to 3-month follow-up; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; t-value on group differences in change = -2.05 — degrees of freedom = 327
Statistical Analysis 3: Comparison: Sham rTMS vs Active rTMS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Comparison of differences between rTMS+CPT and sham+CPT groups in change Clinical Administered Post-Traumatic Scale Total Severity Scores from baseline to 6-month follow-up; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; t-value on group differences in change = -2.01 — degrees of freedom = 327

2. Secondary Outcome: Changes in ERP/CAPS Cluster Scores Signals From Pre-Treatment to Post-Treatment
Description: The secondary outcome measures will be a) the ERP measures of P3a amplitude for hyperarousal to combat threatening stimuli will be compared from post- to pre-treatment b) the total CAPS scores from pre-treatment and post-treatment will be compared.
Time Frame: Outcomes will be assessed at baseline and 6-month follow-up
Population: Sixty participants (6 female) of the 103 completed the study protocol and returned for 6-month follow-up evaluation; the data from those 60 veterans were analyzed and reported.
Measure: Mean (Standard Deviation); unit: micro-volts
Arm/Group | Sham rTMS | Active rTMS
Number analyzed (Participants) | 28 | 32
micro-volts | -1.2754 (3.095) | -0.6088 (2.278)
Statistical Analysis 1: Comparison: Sham rTMS vs Active rTMS; Null hypothesis test of differences in N2 micro-volt change from baseline to 6-month followup; Test type: Superiority; p = .3422, t-test, 2 sided — It is not adjusted for multiple comparisons; degrees of freedom = 58; Mean Difference (Final Values) = -0.666, 1.422% CI 2-sided [-0.7548 to 2.088], Standard Deviation 0.7101 — mean change from baseline to 6-month follow-up, rTMS Active - rTMS Sham
Statistical Analysis 2: Comparison: Sham rTMS vs Active rTMS; The analysis examined the association between change in PTSD symptoms from baseline to 6-month follow-up and the change in N2 amplitude to the threatening stimulus from baseline to 6-month follow-up; Test type: Other — The analysis examined correlations in change in N2 and PTSD symptoms; p = 0.02, Regression, Linear — Not adjusted; Slope = -.30; Correlations for the individual groups were active rTMS r(28)=-.373 and sham rTMS r(32)=-.296

ADVERSE EVENTS:
Time Frame: 10 months
Description: Two participants assigned to receive rTMS and one participant assigned to receive sham rTMS reported headaches and requested termination of the rTMS portion of the therapy.
Arm/Group | Sham rTMS | Active rTMS
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/54
Other Adverse Events (participants affected / at risk) | 1/49 | 2/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham rTMS (N=49) | Active rTMS (N=54)
Headache (General disorders) | 1 (1) | 2 (2) — Two participants assigned to receive rTMS and one participant assigned to receive sham rTMS reported headaches and requested termination of the rTMS portion of the therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No